CLINICAL TRIAL: NCT01586897
Title: The Medication Metronome Project
Brief Title: The Medication Metronome Project - Study to Facilitate Follow-up Testing Resulting From Prescribed Medications to Improve Patient Safety and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Atlas, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R18HS018648 (AHRQ)
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemia
Keywords: health information technology; primary care; visit-independent; medication monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of Medication Metronome (Experimental): Providers allocated to intervention will automatically see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipidemia will initiate the follow-up result monitoring, patient outreach, and PCP reminders that constitute the Medication Metronome system.
  Interventions: Device: Medication Metronome
- Usual Care (Active Comparator): PCPs allocated to the control arm will continue with usual care practices for laboratory monitoring.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Medication Metronome — Providers allocated to intervention will see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipidemia will initiate the follow-up result monitoring, patient outreach, and PCP reminders that constitute the Medication Metronome system.
  Arms: Use of Medication Metronome
Other: Usual Care
  Arms: Usual Care

SUMMARY:
This project tests a model of chronic disease medication management in which the decision to initiate or adjust medical therapy is directly linked to a sequence of subsequent clinical actions (e.g. monitoring for adverse drug events, assessing response to therapy, changing medication dose) performed independently of the office visit. The investigators hypothesize that establishing a visit-independent, health information technology (IT) supported cycle of laboratory monitoring and iterative medication dose adjustment will result in more effective chronic disease care.

DETAILED DESCRIPTION:
To implement a new model of chronic disease management, we will build on our existing electronic health record and integrated data systems to develop an advanced health IT application called the "Medication Metronome" to enable providers to schedule future laboratory tests related to a specific set of medications (for glycemic, cholesterol, and blood pressure management). As these lab test dates become due, the Medication Metronome system will remind patients via letter and inform providers when the tests remain "missing." The goal of this intervention is to implement an efficient, visit-independent system to ensure that patients are rapidly and safely brought to evidence-based treatment goals and to prevent delays in planned laboratory monitoring. This study has the following aims:

Aim 1: To develop the Medication Metronome system. This work involves health IT development and evaluation of design prototypes to create a system that supports timely medication intensification, improves safety, and meets both patient and provider needs.

Aim 2: To conduct a randomized controlled trial of the Medication Metronome system. We will use three target chronic conditions to test different elements of the system. We hypothesize that use of the Medication Metronome system will lead to:

H2a. More effective HbA1c control among patients with type 2 diabetes prescribed hypoglycemic medicines; H2b. Safer medication management among patients with hypertension prescribed thiazide diuretics, angiotensin converting enzyme inhibitors, or angiotensin II receptor blockers; H2c. Both more effective LDL-cholesterol control and safer monitoring for hepatitis among patients with hyperlipidemia prescribed HMG-CoA reductase inhibitors.

Aim 3: To evaluate the impact of the Medication Metronome visit-independent care model on the content of office-based visits. Time spent addressing different clinical care domains will be assessed using audiotape-based content analysis in a subset of selected office visits.

Summary: We will implement, and rigorously evaluate a health IT-supported model of visit-independent medication management designed to enable safer and more effective chronic disease care. We will also carefully investigate the impact of this system on primary care visits. The broader goal of this work is to support health delivery redesign that fosters patient-centered primary care by combining visit-independent medication management with more productive visit-based patient-provider interactions.

ELIGIBILITY:
Inclusion Criteria:

* All primary care physicians from participating practices will be eligible to participate in the study.

  * Patients Eligible for Analysis: The primary unit of analysis will be prescribed medicine, grouped with patient and within prescribing PCP. Three potentially overlapping medication-based cohorts will be defined: 1) Patients prescribed any hypoglycemic agents, 2) Patients prescribed thiazide diuretics, ACE-Is, or ARBs, and 3) Patients prescribed statins. Based on this design, individual patients may contribute to more than one medication analytic cohort.

Exclusion Criteria:

* Patients Excluded from Analysis: Patients who are subsequently identified as having died during the course of the study intervention using the Social Security Death Index, to have left the MGH system, or to have changed PCPs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Atlas, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary Care Physicians were recruited and randomized to intervention or control arms, but data were collected and analyzed for the patients of the Primary Care Physicians.
Groups:
- Use of Medication Metronome: Medication Metronome: Providers allocated to intervention will see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipid.
  26 Primary Care Physicians were randomized to "Use of Medication Metronome" with 2049 patients analyzed.
- Usual Care: PCPs allocated to the control arm will continue with usual care practices for laboratory monitoring.
  Usual Care
  26 Primary Care Physicians randomized to Usual Care, with 1606 patients analyzed.
Period: Overall Study
Arm/Group | Use of Medication Metronome | Usual Care
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Use of Medication Metronome: Medication Metronome: PCPs allocated to intervention will see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipid.
  While PCPs were randomized, analyses were at the patient level. Characteristics presented represent eligible patients of randomized PCPs.
- Usual Care: PCPs allocated to the control arm will continue with usual care practices for laboratory monitoring.
  Usual Care
  While PCPs were randomized, analyses were at the patient level. Characteristics presented represent eligible patients of randomized PCPs.
- Total: Total of all reporting groups
Arm/Group | Use of Medication Metronome | Usual Care | Total
Number analyzed (Participants) | 2049 | 1606 | 3655
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (13.1) | 65.7 (12.8) | 65.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 979 | 850 | 1829
  Male | 1070 | 756 | 1826

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Outcome - LDL
Description: Percentage of follow-up time (from initial prescription to final laboratory result available during the 18-month study period) that a patient is at or below risk factor goal for LDL(LDL-cholesterol ≤ 130 mg/dL for patients without cardiovascular risk and ≤ 100 mg/dl for patients with cardiovascular risk).
Time Frame: 1 year
Population: Patients prescribed statins during the study period
Measure: Mean (Standard Deviation); unit: percentage of time spent at goal
Groups:
- Use of Medication Metronome: Medication Metronome: Providers allocated to intervention will see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipid
- Usual Care: PCPs allocated to the control arm will continue with usual care practices for laboratory monitoring.
  Usual Care
Arm/Group | Use of Medication Metronome | Usual Care
Number analyzed (Participants) | 953 | 703
percentage of time spent at goal | 57.9 (44.4) | 54.8 (46.2)

2. Primary Outcome: Primary Effectiveness Outcome - A1c
Description: Percentage of follow-up time (from initial prescription to final laboratory result available during the 18-month study period) that a patient is at or below risk factor goal for HbA1c(HbA1c ≤ 7.0%).
Time Frame: 1 year
Population: Patients prescribed oral medications for diabetes control during the study period
Measure: Mean (Standard Deviation); unit: percentage of time spent at goal
Arm/Group | Use of Medication Metronome | Usual Care
Number analyzed (Participants) | 318 | 300
percentage of time spent at goal | 32.5 (43.2) | 34.3 (42.5)

3. Primary Outcome: Medication Safety Monitoring - Statins
Description: Percentage of laboratory tests (liver function tests after a new statin prescription or a change in statin dose) that have been measured within 4 weeks following prescription. Treatment guidelines for prescription of statins recommend follow-up liver function testing. We chose 4-weeks following the prescription to represent successful safety monitoring.
Time Frame: Within 4 weeks following prescription
Population: Patients prescribed statins
Measure: Number; unit: percentage of tests within 4 weeks
Arm/Group | Use of Medication Metronome | Usual Care
Number analyzed (Participants) | 1134 | 699
percentage of tests within 4 weeks | 6.7 | 8.6

4. Primary Outcome: Medication Safety Monitoring - Metformin
Description: Percentage of renal function laboratory tests that have been measured within 4-weeks following prescription. Treatment guidelines for prescription of metformin recommend renal function testing. We chose 4- weeks following the prescription to represent successful safety monitoring.
Time Frame: Within 4 weeks following prescription
Population: Patients prescribed metformin
Measure: Number; unit: percentage of tests within 4 weeks
Arm/Group | Use of Medication Metronome | Usual Care
Number analyzed (Participants) | 445 | 425
percentage of tests within 4 weeks | 13.7 | 16.2

5. Primary Outcome: Medication Safety Monitoring - ACE/ARB, Thiazide
Description: Percentage of laboratory tests (potassium for thiazides, renal/potassium for ACE/ARBs that have been measured within 4-weeks following prescription. Treatment guidelines for prescription of ACE/ARBs recommend renal/potassium testing and potassium testing for prescription of thiazides. We chose 4-weeks following the prescription to represent successful safety monitoring.
Time Frame: Within 4 weeks following prescription
Population: Patients prescribed ACE/ARB, thiazide
Measure: Number; unit: percentage of tests within 4 weeks
Arm/Group | Use of Medication Metronome | Usual Care
Number analyzed (Participants) | 1411 | 1296
percentage of tests within 4 weeks | 26.9 | 24.0

ADVERSE EVENTS:
Groups:
- Use of Medication Metronome - PCPs: Medication Metronome: Providers allocated to intervention will see an additional feature when logging on to their electronic health record medication prescription interface that enables them to schedule future laboratory testing for the pre-defined subset of study-specific medications. New prescription or dose adjustment by the PCP of one of these pre-specified medications used to treat type 2 diabetes, hypertension, or hyperlipidemia.
- Usual Care - PCPs: PCPs allocated to the control arm will continue with usual care practices for laboratory monitoring.
  Usual Care
- Use of Medication Metronome - Patients: Patients of PCPs allocated to the "Use of Medication Metronome" were eligible for our outcomes if prescribed a new study medication or if they experienced a dose change of a study medication.
- Usual Care - Patients: Patients of PCPs allocated to "Usual Care" were eligible for our outcomes if prescribed a new study medication or if they experienced a dose change of a study medication.
Arm/Group | Use of Medication Metronome - PCPs | Usual Care - PCPs | Use of Medication Metronome - Patients | Usual Care - Patients
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/2049 | 0/1606
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/2049 | 0/1606

LIMITATIONS AND CAVEATS:
Study participants did not embrace this method of non-visit based care, with only 660 medication prescriptions using the Medication Metronome ordering option (21% of possible orders).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No